CLINICAL TRIAL: NCT05780515
Title: A Single-Arm, Phase 1b, Open-Label Study to Assess the Safety, Tolerability, and Pharmacodynamics of Repeat-Doses of Subcutaneous ANX009 With Standard of Care Therapy in Adult Participants With Lupus Nephritis
Brief Title: A Study of ANX009 in Adult Participants With Lupus Nephritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Annexon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANX009-LN-01
Record Dates: First submitted 2023-03-10; First posted 2023-03-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Immunoglobulin G; Immunoglobulin Fab Fragments

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ANX009 (Experimental): Participants will receive repeat doses of ANX009 administered by subcutaneous (SC) infusion 3 times weekly during the approximate 3-week intervention period.
  Interventions: Biological: ANX009

INTERVENTIONS:
Biological: ANX009 — ANX009 will be administered per schedule specified in the arm description.
  Other Names: Recombinant humanized immunoglobulin G1 (IgG1) Fab

SUMMARY:
The main purpose of this study is to determine the safety and tolerability of repeat doses of ANX009 in participants with lupus nephritis (LN).

DETAILED DESCRIPTION:
All participants may continue to receive stable background standard of care therapy for LN and systemic lupus erythematosus (SLE) as permitted by the protocol (for example, mycophenolate mofetil [MMF], azathioprine, antimalarials, glucocorticoids, cyclosporin, voclosporin, tacrolimus, angiotensin converting enzyme [ACE] inhibitors, angiotensin receptor blockers [ARBs]).

ELIGIBILITY:
Key Inclusion Criteria:

* Participants who have a diagnosis of SLE according to European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) 2019 Criteria
* Has a history of International Society of Nephrology/Renal Pathology Society (ISN/RPS) Class III or IV with or without Class V glomerulonephritis on renal biopsy within 24 months prior to screening or as performed during screening.
* Has proteinuria level between ≥0.5 to 3.0 grams (g)/g/day assessed via urine protein to creatine ratio (UPCR) during screening.
* Has evidence of classical complement activation at screening
* Has a history of receiving one or more standard therapies for LN

Key Exclusion Criteria:

* Has a history of ISN/RPS Class VI or isolated Class V (without co-existent/predominant Class III or IV glomerulonephritis) glomerulonephritis on renal biopsy.
* Has severe kidney disease defined as eGFR of <30 milliliters (mL)/minute/1.73 square meter (m^2) or end-stage renal disease (ESRD) requiring dialysis or kidney transplantation.
* Has a concurrent systemic autoimmune disease that may confound study assessments other than SLE, LN, or cutaneous lupus erythematosus.

NOTE: Other inclusion and/or exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | Baseline (Week 1) up to Week 15

SECONDARY OUTCOMES:
Change From Baseline in Free Complement Component 1q (C1q) Concentrations in Serum Over Time | Baseline (Week 1), up to Day 31
Change From Baseline in Complement Factor C4 Concentration and its Activation Product (Complement Component 4d [C4d]) in Plasma Over Time | Baseline (Week 1), up to End of Study (up to Week 15)

CONTACTS AND LOCATIONS:
Overall Officials: Annexon Director Global Clinical Operations, Study Director — Annexon, Inc.
Locations (7):
- Philippines (4):
  - Annexon Investigational Site 203, Angeles City
  - Annexon Investigational Site 204, Iloilo City
  - Annexon Investigational Site 201, Manila
  - Annexon Investigational Site 202, Quezon City
- Taiwan (3):
  - Annexon Investigational Site 101, Taichung
  - Annexon Investigational Site 102, Taipei
  - Annexon Investigational Site 103, Taoyuan